CLINICAL TRIAL: NCT06416761
Title: The Genetic Contribution to Progression of Kidney Disease
Brief Title: Genetics in the Progression of Nephropathies
Status: Recruiting | Type: Observational
Sponsor: Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Chiara Lanzani, Clinical Assistant, Ospedale San Raffaele
Other Study IDs: GenNefro01
Record Dates: First submitted 2024-05-11; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: AKI; CKD; Ckd-Mbd; CKD (Chronic Kidney Disease) Stage 5D; ADPKD; Hypertension; Hematologic Malignancy; Bone Marrow Transplant Complications
Keywords: genetic in hypertensive kidney disease; salt intake in BP control and CKD progression; genetic in CKD; endogenous Ouabain as marker of AKI; protein intake restriction in CKD progression; hypertension in allogenic bone marrow transplantation
MeSH Terms: conditions — Chronic Kidney Disease-Mineral and Bone Disorder; Renal Insufficiency, Chronic; Polycystic Kidney, Autosomal Dominant; Hypertension; Hematologic Neoplasms | interventions — Polymorphism, Genetic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — blood , urine and sample of renal tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with acute or chronic nephropathy: 1. Patients with chronic nephropathies
  2. Patients with acute nephropathy
  3. Patients with nephrectomy
  4. Candidate Patients to major surgery
  5. Patients with decompensated heart failure undergoing either medical or surgical therapy
  6. Acute critically ill patients (e.g sepsis, post-operative)
  7. Patients with hypertension
  8. Patients with hematologic cancer exposed to chemotherapeutic agents or undergoing allogeneic bone marrow transplantation.
  9. Long-term surviving patients who received bone marrow transplantation.
  Interventions: Genetic: genetic polymorphisms

INTERVENTIONS:
Genetic: genetic polymorphisms

SUMMARY:
This study evaluates the role of genetic in the development and progression of different nephropaties with particular attention to:

* AKI
* CKD
* Hypertension
* ADPKD
* CKD-MBD
* Patients with decompensated heart failure undergoing either medical or surgery therapy
* Patients with hematologic cancer exposed to chemotherapeutic agents or undergoing allogeneic bone marrow transplantation
* glomerular diseases

DETAILED DESCRIPTION:
Background: In the past ten years there's been a progressive increase in the prevalence of CKD and consequently in the number of dialysed patients (~4% per year) in Italy. This is probably due to the increasingly ageing population and incidence of CV disease (cf. Lombardy Register). To date, diabetes and CV disease are the most common cause of end-stage renal disease (ESRD) requiring RRT. Nonetheless, intrinsic renal diseases still remain an important cause of CKD. In the past few years, various environmental factors have been identified that affect the clinical progression of kidney disease: blood pressure control, lipid and glycemic profile (expecially in the setting of diabetic nephropaty), uric acid level and acid-base homeostasis. Recently, there have been found some genes responsible for monogenic hereditary diseases such as ADPKD (PKD1 e PKD2) and Alport syndrome (COL4A3/COL4A4/COL4A5). It is known that there's an important phenotypic heterogeneity among different patients with the same disease even in the same family because of incomplete penetrance [5]. Furthermore, it is well known that familiarity overbear all other risk factors in predicting the development of hypertension and its progression toward CKD. Many scientific findings show the link between some genetic polymorphisms (e.g ACE, adducin) and disease severity or development of various complications. There is now, increasingly scientific evidence that genetic palys an important role even in the development and progression of multifactorial renal disease with both protective or promoting possible pathways. Thus, It would seem that interactions between environmental and genetic factors are responsible for disease phenotypic heterogeneity and its progression.

Aim of the study:

* Extend the knowledge on genetic modifiers involved in disease progression to better classify patients in homogeneous groups based on aetiology and concomitant risk factors. According to the underlying pathology, patients will be assessed either alone or with their family to evaluate the phenotypic heterogeneity.
* Evaluate the role of drugs that targets genetic or environmental factors.
* Assess the role of gentic background in the development of CV complications in CKD patients undergoing dyalisis.
* Assess the role of immature progenitor cells in the progression of kidney disease.
* Evaluate the role of endogenous Ouabain to identify at increased risk for AKI: 1) Postoperative patients. 2) patients with decompensated heart failure undergoing surgery or PCI. 3) patients with severe hypovolemic shock due to either cardiologic causes (e.g AMI) or from other causes (e.g sepsis, hypertensive crisis) 4) patients with hematologic cancer exposed to chemotherapeutic agents or undergoing allogeneic bone marrow transplantation.
* Identify the presence of genetic modifiers influencing the development and progression of CKD.
* Evaluate the role of genetic polymorphism in the transition from hypertension to kidney disease.
* Assess the role of salt intake in BP control and CKD progression either alone or in the presence of genetic modifiers.
* Evaluate the role of protein intake restriction in CKD progression eitehr alone or in the presence of genetic modifiers.
* Identify cortical bone lesions in CKD
* Assess the role of genetic, nutritional and biochemical factors involved in the cortical bone development
* Evaluate the role of genetic in the development of hypertension in patients who received allogenic bone marrow transplantation.

The genetic polymorphisms that will be considered, based on current knowledge are:

* Alpha, beta, gamma Adducin (ADD1, ADD2, ADD3),
* Renin Angiotensin System (RAAS),
* Glomerular proteins: nephrine, podocin, cadherin.
* Renal tubular transport systems (Na-Cl cotransport, Na channel, lithium, Cl channel, K channel, Ca channel, Amino Acids, specialized tubular transporters ouabain, drugs, digoxin, aquaporins, ANP, BNP).
* Genes linked to the metabolism and function of endogenous ouabain (eg LSS) and Klotho (eg KL).
* Polycystin 1, polycystin 2 (PKD1 and PKD2), uromodulline, S. di Alport (COL4A3/COL4A4/COL4A5)

For the study of any further genetic polymorphisms, additional amendments to this research protocol will be formulated.

ELIGIBILITY:
Inclusion Criteria:

. presence of specific renal disease

Exclusion Criteria:

* to be evaluated in the different sub-protocols

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will evaluate different groups of adult patients:
  1. Patients with chronic nephropathy
  2. Patients with acute nephropathy
  3. Patients with nephrectomy
  4. Candidate Patients to major surgery
  5. Patients with decompensated heart failure undergoing either medical or surgical therapy
  6. Acute critically ill patients (e.g sepsis, post-operative)
  7. Patients with hypertension
  8. Patients with hematologic cancer exposed to chemotherapeutic agents or undergoing allogeneic bone marrow transplantation.
  9. Long-term surviving patients who received bone marrow transplantation.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2006-05-19 (Actual); Primary Completion 2040-05-19 (Estimated); Study Completion 2041-05-19 (Estimated)

PRIMARY OUTCOMES:
difference in glomerular filtration rate according to genetic profile | from days to 35 years
  eGFR value

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy